CLINICAL TRIAL: NCT00045110
Title: A Phase I/II Trial of OSI-774 in Patients With Recurrent Malignant Gliomas and Malignant Gliomas Post Radiation Therapy
Brief Title: Erlotinib in Treating Patients With Recurrent Malignant Glioma or Recurrent or Progressive Meningioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02490; NCI-2012-02490 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-03-C-0114; CDR0000256358; NABTC-01-03 (Other: North American Brain Tumor Consortium); NABTC-01-03 (Other: CTEP); U01CA062399 (NIH); NCT00055276 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Grade I Meningioma; Adult Grade II Meningioma; Adult Grade III Meningioma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Meningioma; Brain Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Phase I: Patients concurrently receiving EIAEDs receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  erlotinib hydrochloride given orally
  Other: pharmacological study.
  Interventions: Drug: erlotinib hydrochloride; Other: pharmacological study
- Phase 2 recurrent malignant gliomas and nonprogressive GBM (Experimental): Phase II: Patients not concurrently receiving EIAEDs are treated with erlotinib as above at a predetermined dose (150mg/day.
  patients requiring surgery treated 7 days prior to tumor removal (150mg/day)
  PK analysis and effects of erlotinib on epidermal growth factor receptor (EGFR)
  erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: erlotinib hydrochloride — given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — correlative studies
  Arms: Phase 2 recurrent malignant gliomas and nonprogressive GBM
Other: pharmacological study — correlative studies

SUMMARY:
Phase I/II trial to study the effectiveness of erlotinib in treating patients who have recurrent malignant glioma or recurrent or progressive meningioma. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase 1 I. Determine the maximum tolerated dose of erlotinib in patients with recurrent malignant glioma or recurrent or progressive meningioma.

II. Determine the safety profile of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients.

Phase 2 I. Determine the 6-month progression-free survival (recurrent malignant glioma) II.12-month survival of patients treated with this drug (stable glioblastoma post radiation therapy)

Phase 2 - Secondary Recurrent Malignant Glioma I. Objective Tumor Response rate associated with erlotinib therapy in recurrent or progressive malignant glioma.

III. 12-month survival of patients treated with this drug Determine the safety profile of this drug in these patients. IV.. Determine the pharmacokinetics of this drug in these patients

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to study phase (I vs II), concurrent enzyme-inducing antiepileptic drugs (EIAEDs) (yes vs no), histology (recurrent GBM vs recurrent anaplastic glioma vs recurrent meningioma vs stable GBM), preoperative candidacy (yes vs no), and concurrent steroids (yes vs no).

Phase I: Patients concurrently receiving EIAEDs receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Phase II: Once the MTD is determined, additional patients concurrently receiving EIAEDs are treated with erlotinib as above at the phase II dose. Patients not concurrently receiving EIAEDs are treated with erlotinib as above at a predetermined dose.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses:

  * Histologically confirmed intracranial malignant glioma

    * Glioblastoma multiforme (GBM), anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed oligoastrocytoma, or malignant astrocytoma not otherwise specified
    * Original histology of low-grade glioma allowed provided a subsequent histology of malignant glioma is confirmed
  * Histologically or radiographically confirmed recurrent or progressive benign or malignant meningioma
* Progressive disease or tumor recurrence on MRI or CT scan

  * Phase I: No more than 3 prior relapses and no more than 2 prior chemotherapy* or biologic therapy regimens
  * Phase II: No more than 2 prior relapses and no more than 2 prior chemotherapy* or biologic therapy regimens
* Patients with progressive disease must have failed prior radiotherapy* that was completed at least 4 weeks ago

  * Patients with progressive disease between 4 and 12 weeks after completion of external beam radiotherapy must have clear evidence of progression on MRI
  * Patients with GBM who have completed external beam radiotherapy and do not show progression are eligible
  * Patients with progressive disease after interstitial brachytherapy or stereotactic radiosurgery must have confirmed true progression rather than radiation necrosis based upon positron-emission tomography, thallium scanning, MRI, or surgical documentation
* Measurable or evaluable disease
* Performance status - Karnofsky 60-100%
* More than 8 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 mg/dL (transfusion allowed)
* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT less than 1.5 times ULN
* Creatinine less than 1.5 mg/dL
* None of the following ophthalmic abnormalities:

  * Abnormalities of the cornea (e.g., dry eye syndrome or Sjögren's syndrome)
  * Congenital abnormality (e.g., Fuch's dystrophy)
  * Abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
  * Abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Patients found to have dry eyes on examination but have an otherwise normal examination allowed
* No active infection
* No other serious concurrent medical illness
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other disease that would obscure toxicity or dangerously alter drug metabolism
* No significant medical illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 12 weeks after study participation
* See Disease Characteristics
* At least 1 week since prior thalidomide
* At least 1 week since prior interferon
* At least 4 weeks since prior SU5416 or other experimental biologic agents
* See Disease Characteristics
* No prior chemotherapy (including polifeprosan 20 with carmustine implant [Gliadel wafers]) for patients with stable GBM
* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 6 weeks since prior nitrosoureas
* At least 1 week since prior tamoxifen
* See Disease Characteristics
* Recovered from prior radiotherapy
* No more than 6 weeks since prior external beam radiotherapy for patients with GBM without evidence of progression
* Recovered from prior surgery
* Recovered from prior therapy
* At least 1 week since prior noncytotoxic agents (e.g., isotretinoin) except radiosensitizers
* At least 4 weeks since prior cytotoxic therapy
* At least 4 weeks since prior tipifarnib or imatinib mesylate
* No prior erlotinib or other epidermal growth factor receptor inhibitors
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2002-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Abrey, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (7):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - National Cancer Institute Neuro-Oncology Branch, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raizer JJ, Abrey LE, Lassman AB, Chang SM, Lamborn KR, Kuhn JG, Yung WK, Gilbert MR, Aldape KD, Wen PY, Fine HA, Mehta M, Deangelis LM, Lieberman F, Cloughesy TF, Robins HI, Dancey J, Prados MD; North American Brain Tumor Consortium. A phase I trial of erlotinib in patients with nonprogressive glioblastoma multiforme postradiation therapy, and recurrent malignant gliomas and meningiomas. Neuro Oncol. 2010 Jan;12(1):87-94. doi: 10.1093/neuonc/nop017. Epub 2009 Dec 14. PMID 20150371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled between August 15, 2002 and August 18, 2005. Patient recruited from outpatient oncology centers.
Groups:
- Phase 1 Dose Escalation: Phase I: Patients concurrently receiving EIAEDs receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis.
- Phase 2 - Recurrent Malignant Glioma: Phase II: Once the MTD is determined, additional patients concurrently receiving EIAEDs are treated with erlotinib as above at the phase II dose.
  Patients not concurrently receiving EIAEDs are treated with erlotinib as above at a predetermined dose.
  patients requiring surgery were treated 7 days prior to tumor removal; PK analysis and effects of erlotinib on epidermal growth factor receptor (EGFR)
  erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis.
- Phase 2 - Newly Diagnosed GBM Post RT: Patients with GBM with newly diagnosed disease following Radiation (RT) started erlotinib no more than 6 weeks from the completion of RT. Temozolomide or other adjuvant chemotherapy not allowed while on erotinib
Period: 100mg Phase 1 Dose Escalalation
Arm/Group | Phase 1 Dose Escalation | Phase 2 - Recurrent Malignant Glioma | Phase 2 - Newly Diagnosed GBM Post RT
Started | 6 | 59 | 45
Completed | 6 | 53 | 43
Not Completed | 0 | 6 | 2
Not completed — did not initiate treatment | 0 | 2 | 1
Not completed — prior treatment history | 0 | 4 | 0
Not completed — ineligible histology | 0 | 0 | 1
Period: 200mg Phase 1 Dose Escalation
Arm/Group | Phase 1 Dose Escalation | Phase 2 - Recurrent Malignant Glioma | Phase 2 - Newly Diagnosed GBM Post RT
Started | 4 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 0 | 0 | 0
Period: 275mg Phase 1 Dose Escalation
Arm/Group | Phase 1 Dose Escalation | Phase 2 - Recurrent Malignant Glioma | Phase 2 - Newly Diagnosed GBM Post RT
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: 400mg Phase 1 Dose Escalation
Arm/Group | Phase 1 Dose Escalation | Phase 2 - Recurrent Malignant Glioma | Phase 2 - Newly Diagnosed GBM Post RT
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: 525mg Phase 1 Dose Escalation
Arm/Group | Phase 1 Dose Escalation | Phase 2 - Recurrent Malignant Glioma | Phase 2 - Newly Diagnosed GBM Post RT
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: 650mg Phase 1 Dose Escalation
Arm/Group | Phase 1 Dose Escalation | Phase 2 - Recurrent Malignant Glioma | Phase 2 - Newly Diagnosed GBM Post RT
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: 775mg Dose Escalation
Arm/Group | Phase 1 Dose Escalation | Phase 2 - Recurrent Malignant Glioma | Phase 2 - Newly Diagnosed GBM Post RT
Started | 7 | 0 | 0
Completed | 7 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: enrolled between 8/2002 and 8/2005. All recruited from outpatient setting.
Groups:
- Phase 2 w/ Recurrent Malignant Glioma: Phase II: Patients not concurrently receiving EIAEDs are treated with erlotinib at a predetermined dose (150mg/day).
  Patients requiring surgery were treated 7 days prior to tumor removal PK analysis and effects of erlotinib on epidermal growth factor receptor (EGFR) erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis
- Phase 2 Newly Diagnosed GBM Post RT: Phase II: Patients not concurrently receiving EIAEDs are treated with erlotinib as above at a predetermined dose. (150mg/day)
  erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation | Phase 2 w/ Recurrent Malignant Glioma | Phase 2 Newly Diagnosed GBM Post RT | Total
Number analyzed (Participants) | 32 | 59 | 45 | 136
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 76] | 54 [29 to 78] | 52 [19 to 72] | 52 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 25 | 10 | 47
  Male | 20 | 34 | 35 | 89
Histology [Number; unit: participants]
  Glioblastoma | 21 | 42 | 44 | 107
  Anaplastic Astrocytoma | 8 | 14 | 1 | 23
  Anaplastic oligodendroglioma | 2 | 1 | 0 | 3
  Atypical meningioma | 1 | 0 | 0 | 1
  Pleomorphic Xanthoastrocytoma | 0 | 1 | 0 | 1
  Oligodendroglioma | 0 | 1 | 0 | 1
Prior Radiation Treatment [Number; unit: participants]
  Yes | 32 | 55 | 45 | 132
  No | 0 | 4 | 0 | 4
Prior Number of Chemotherapy Regimens [Number; unit: participants]
  0 treatments | 3 | 4 | 0 | 7
  1 treatment | 13 | 31 | 45 | 89
  2 treatments | 14 | 21 | 0 | 35
  3 treatments | 2 | 3 | 0 | 5
Karnofsky Performance Status Scale [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 90 [60 to 100] | 80 [60 to 100] | 90 [60 to 100] | 80 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicity (DLT) Each Dose Level Phase I
Description: DLT Definition: any grade 3 thrombocytopenia and grade 4 anemia and neutropenia; any non-hematologic grade 3 toxicity; failure to recover from toxicities to be eligible for re-treatment with erlotinib within 2 weeks of the last dose of erlotinib.
Time Frame: 28 days
Population: Patients were eligible if they had recurrent disease or if they were newly diagnosed post RT and did NOT have tumor progression (nonprogression glioblastoma) on Enzyme-inducing Antiepileptic Drugs
Measure: Number; unit: dose limiting toxicities
Groups:
- Phase 1 Dose Escalation: Phase I: Patients concurrently receiving EIAEDs ( on Enzyme-inducing Antiepileptic Drugs ) receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined.
  The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Other: pharmacological study, laboratory biomarker analysis.
Arm/Group | Phase 1 Dose Escalation
Number analyzed (Participants) | 32
dose limiting toxicities
  Dose 150mg (Rash): number analyzed (Participants) | 6
  Dose 150mg (Rash) | 1
  Dose 200mg: number analyzed (Participants) | 3
  Dose 200mg | 0
  Dose 275mg: number analyzed (Participants) | 3
  Dose 275mg | 0
  Dose 400mg: number analyzed (Participants) | 3
  Dose 400mg | 0
  Dose 525mg: number analyzed (Participants) | 3
  Dose 525mg | 0
  Dose 650mg (DVT/PE): number analyzed (Participants) | 6
  Dose 650mg (DVT/PE) | 1
  Dose 775mg (Rash [2]): number analyzed (Participants) | 6
  Dose 775mg (Rash [2]) | 2

2. Primary Outcome: Define Maximum Tolerated Dose (MTD) of Erlotinib by Phase 1 Cohorts
Description: standard 3+3 dose escalation design 3 patients in each dose level, observed for 28 days before enrollment to next level. if none of the patients experienced DLT dose escalated, if 1 of 3 experienced DLT 3 more enrolled at that level, if none of the 3 additional pts had DLT escalate to next level, if one or more of the additional pts experienced DLT, the MTD was exceeded and 3 more patients were treated at the next lower dose (if only 3 pts treated at the lower dose). The MTD is the dose at which 0/3 or 1/6 patients have experienced a DLT with the next higher dose having at least 2/3 or 2/6 patients encountering DLT.
Time Frame: cycle 1 - 28 days
Population: Cohorts/dose levels: 150mg; 200mg; 275mg; 400mg; 525mg; 650mg; 775mg patients on Enzyme-inducing Antiepileptic Drugs
Measure: Number; unit: mg
Groups:
- Phase 1 Dose Escalation: Phase I: Patients concurrently receiving EIAEDs ( on Enzyme-inducing Antiepileptic Drugs) receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined.
  The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Other: pharmacological study, laboratory biomarker analysis.
Arm/Group | Phase 1 Dose Escalation
Number analyzed (Participants) | 32
mg | 650

3. Primary Outcome: 6 Months Progression-free Survival in Recurrent Malignant Gliomas (Phase II)
Description: Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over BL if no decrease), OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months
Population: 38 Glioblastoma, 15 anaplastic gliomas not receiving Enzyme-inducing Antiepileptic Drugs
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Recurrent Malignant Gliomas: Phase II: Patients not concurrently receiving EIAEDs are treated with erlotinib as above at a predetermined dose.
  patients requiring surgery were treated 7 days prior to tumor removal
  PK analysis and effects of erlotinib on epidermal growth factor receptor (EGFR)
  erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis.
  erlotinib hydrochloride: given orally
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
Arm/Group | Phase 2 Recurrent Malignant Gliomas
Number analyzed (Participants) | 53
Participants
  Recurrent GBM | 2
  Recurrent Anaplastic Glioma | 14

4. Secondary Outcome: Percent of Participants With a Grade 3 or 4 Adverse Events Phase 1
Description: CTCAE
Time Frame: 1 year
Population: During Cycle 1 only grade 3 severity; patients on Enzyme-inducing Antiepileptic Drugs
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Dose Escalation: Phase I: Patients concurrently receiving EIAEDs (on Enzyme-inducing Antiepileptic Drugs) receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined.
  The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Other: pharmacological study, laboratory biomarker analysis..
  erlotinib hydrochloride: given orally
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
Arm/Group | Phase 1 Dose Escalation
Number analyzed (Participants) | 32
Participants | 4

5. Secondary Outcome: 1 Year Survival - Phase II Newly Diagnosed GBM Post RT
Description: 12 month survival for newly diagnosed stable GBM post RT treated with erlotinib post RT
Time Frame: At 1 year
Population: not receiving Enzyme-inducing Antiepileptic Drugs; stable glioblastoma after RT
Measure: Number; unit: % of participants
Arm/Group | Phase 2 Newly Diagnosed GBM Post RT
Number analyzed (Participants) | 43
% of participants | 57

6. Secondary Outcome: Overall Survival Newly Diagnosed GBM Post RT
Description: Overall Survival defined as Time from Start of treatment to time of death due to any cause
Time Frame: 2 years
Population: not receiving Enzyme-inducing Antiepileptic Drugs, glioblastoma stable after RT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Newly Diagnosed GBM Post RT
Number analyzed (Participants) | 45
months | 14 [9 to 17]

7. Secondary Outcome: Response Rate (Complete or Partial Response) Graded Using Modified RECIST Criteria Phase II
Description: Measurable: Bidimensionally measurable lesions w/ clearly defined margins by MRI
  Evaluable: Unidimensionally measurable lesions, masses w/margins not clearly defined.
  Complete Response (CR): Complete disappearance of all measurable/evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients on minimal/no steroids.
  Partial Response (PR): >/= to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. Responders must be on same/decreasing doses of dexamethasone.
  Stable/No Response: Does not qualify for CR, PR, or progression.
  Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over BL if no decrease), OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: At 1 year
Population: recurrent malignant gliomas - anaplastic and glioblastoma
Measure: Number; unit: participants
Arm/Group | Phase 2 Recurrent Malignant Gliomas
Number analyzed (Participants) | 48
participants
  complete response | 1
  Partial response | 1
  stable disease | 5
  Progression | 41

8. Secondary Outcome: Percent of Patients With One or More Grade 3-5 Toxicity Described Based on the CTC Severity Grading Phase II
Description: Summarized by descriptive statistics.
Time Frame: Up to 1 year
Population: drug related events grade 3-5 CTCAE. 5 patients were not evaluable for response/toxicity.
Measure: Number; unit: percent of participants
Groups:
- Phase 2 Recurrent Malignant Gliomas and Stable Disease Post RT: Patients with recurrent malignant gliomas not concurrently receiving EIAEDs treated with erlotinib at a predetermined dose.
  patients requiring surgery were treated 7 days prior to tumor removal
  PK analysis and effects of erlotinib on epidermal growth factor receptor (EGFR)
  erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis.
  erlotinib hydrochloride: given orally
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
Arm/Group | Phase 2 Recurrent Malignant Gliomas and Stable Disease Post RT
Number analyzed (Participants) | 99
percent of participants | 29

9. Secondary Outcome: Time of Peak Plasma Concentration Per Dose Level Phase I (on Anticonvulsants) -
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: baseline, 1,2,4,6,8,12,24h post administration day 1 cycle 1.
Population: tmax=time of peak plasma concentration
Measure: Mean (Standard Deviation); unit: h
Groups:
- Phase 1 Dose Escalation - 150 mg: Phase I: Patients concurrently receiving EIAEDs receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined.
  The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Other: pharmacological study, laboratory biomarker analysis.
- Phase 1 Dose Escalation - 200 mg; Phase 1 Dose Escalation - 275 mg; Phase 1 Dose Escalation - 400 mg; Phase 1 Dose Escalation - 525 mg; Phase 1 Dose Escalation - 650 mg; Phase 1 Dose Escalation - 775 mg: Phase I: Patients concurrently receiving EIAEDs receive oral erlotinib once daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined.
  The MTD is the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
Arm/Group | Phase 1 Dose Escalation - 150 mg | Phase 1 Dose Escalation - 200 mg | Phase 1 Dose Escalation - 275 mg | Phase 1 Dose Escalation - 400 mg | Phase 1 Dose Escalation - 525 mg | Phase 1 Dose Escalation - 650 mg | Phase 1 Dose Escalation - 775 mg
Number analyzed (Participants) | 6 | 4 | 1 | 2 | 2 | 6 | 5
h | 2.3 (1.37) | 2.8 (2.2) | 3.3 (1.2) | 6 (0) | 3.5 (3.54) | 2.2 (0.98) | 2.4 (2.07)

10. Secondary Outcome: Peak Plasma Concentration Per Dose Level Phase I (on Anticonvulsants) -
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: baseline, 1,2,4,6,8,12,24h post administration day 1 cycle 1. One sample on day 8 cycle 1 and day 1 of cycle 2,3 and 5
Population: Cp=peak plasma concentration;
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 Dose Escalation - 150 mg | Phase 1 Dose Escalation - 200 mg | Phase 1 Dose Escalation - 275 mg | Phase 1 Dose Escalation - 400 mg | Phase 1 Dose Escalation - 525 mg | Phase 1 Dose Escalation - 650 mg | Phase 1 Dose Escalation - 775 mg
Number analyzed (Participants) | 6 | 4 | 1 | 2 | 2 | 6 | 5
ng/mL | 603 (160) | 722 (186) | 1075 (308) | 487 (0) | 2327 (1609) | 1351 (441) | 2009 (1133)

11. Secondary Outcome: Estimation of the Area Under the Curve Per Dose Level Phase I (on Anticonvulsants) -
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: baseline, 1,2,4,6,8,12,24h post administration day 1 cycle 1. One sample on day 8 cycle 1 and day 1 of cycle 2,3 and 5
Population: AUC=area under the curve
Measure: Mean (Standard Deviation); unit: ug* h/mL
Arm/Group | Phase 1 Dose Escalation - 150 mg | Phase 1 Dose Escalation - 200 mg | Phase 1 Dose Escalation - 275 mg | Phase 1 Dose Escalation - 400 mg | Phase 1 Dose Escalation - 525 mg | Phase 1 Dose Escalation - 650 mg | Phase 1 Dose Escalation - 775 mg
Number analyzed (Participants) | 6 | 4 | 1 | 2 | 2 | 6 | 5
ug* h/mL | 5.33 (2.04) | 7.28 (2.54) | 13.58 (2.99) | 21.09 (0) | 25.94 (21.6) | 15.77 (7.43) | 18.83 (11.9)

12. Secondary Outcome: Trough Level Per Dose Level Phase I (on Anticonvulsants) -
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: cycle 1 day eight
Population: trough level
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 Dose Escalation - 150 mg | Phase 1 Dose Escalation - 200 mg | Phase 1 Dose Escalation - 275 mg | Phase 1 Dose Escalation - 400 mg | Phase 1 Dose Escalation - 525 mg | Phase 1 Dose Escalation - 650 mg | Phase 1 Dose Escalation - 775 mg
Number analyzed (Participants) | 6 | 4 | 1 | 2 | 2 | 6 | 5
ng/mL | 412 (430) | 227 (82) | 821 (154) | 634 (0) | 1356 (132) | 591 (574) | 942 (775)

13. Secondary Outcome: Peak Plasma Concentration Level for Recurrent Patients Not on Enzyme-inducing Antiepileptic Drugs - Phase 2 - Dose 150mg -
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: baseline, 1,2,4,6,8,12,24h post administration day 1 cycle 1. One sample on day 8 cycle 1 and day 1 of cycle 2,3 and 5
Population: Cpmax =peak plasma concentration;
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2 Recurrent Malignant Gliomas
Number analyzed (Participants) | 76
ng/mL | 872 (399)

14. Secondary Outcome: Time to Peak Plasma Concentration for Recurrent Patients Not on Enzyme-inducing Antiepileptic Drugs - Phase 2 - Dose 150mg -
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: baseline, 1,2,4,6,8,12,24h post administration day 1 cycle 1. One sample on day 8 cycle 1 and day 1 of cycle 2,3 and 5
Population: tmax=time to peak plasma concentration;
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Phase 2 Recurrent Malignant Gliomas
Number analyzed (Participants) | 76
h | 3.0 (1.91)

15. Secondary Outcome: Estimation of Area Under the Curve for Recurrent Patients Not on Enzyme-inducing Antiepileptic Drugs - Phase 2 - Dose 150mg-
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: baseline, 1,2,4,6,8,12,24h post administration day 1 cycle 1. One sample on day 8 cycle 1 and day 1 of cycle 2,3 and 5
Population: AUC=area under the curve;
Measure: Mean (Standard Deviation); unit: ug * h/mL
Arm/Group | Phase 2 Recurrent Malignant Gliomas
Number analyzed (Participants) | 76
ug * h/mL | 11.86 (5.01)

16. Secondary Outcome: Trough Level for Recurrent Patients Not on Enzyme-inducing Antiepileptic Drugs - Phase 2 - Dose 150mg -
Description: plasma concentrations relative to erlotiniab administration and sample time and dose level
Time Frame: One sample on day 8 cycle 1
Population: Cp=peak plasma concentration; tmax=time to Cp; AUC=area under the curve;
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2 Recurrent Malignant Gliomas
Number analyzed (Participants) | 76
ng/mL | 975 (535)

17. Secondary Outcome: Pharmacokinetics (Plasma) Level for Recurrent Patients Not on Enzyme-inducing Antiepileptic Drugs
Description: Drug administered 6 days prior to surgery
Time Frame: Pre-surgery and time of resection
Population: sample 5 and 6 suspected of contamination with blood clot
Measure: Mean (Standard Deviation); unit: plasma concentration ng/mL
Arm/Group | Phase 2 Newly Diagnosed GBM Post RT
Number analyzed (Participants) | 6
plasma concentration ng/mL | 761 (499)

18. Secondary Outcome: Pharmacokinetics (Tissue) Level for Recurrent Patients Not on Enzyme-inducing Antiepileptic Drugs
Description: Drug administered 6 days prior to surgery
Time Frame: Pre-surgery and time of resection
Population: sample 5 and 6 suspected of contamination with blood clot tumor/tissue concentration
Measure: Mean (Standard Deviation); unit: tumor/tissue concentration ng/g dry weig
Arm/Group | Phase 2 Newly Diagnosed GBM Post RT
Number analyzed (Participants) | 6
tumor/tissue concentration ng/g dry weig | 497 (353)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Phase 2 Recurrent Malignant Gliomas and Nonprogressive Gbm: Phase II: Patients not concurrently receiving EIAEDs are treated with erlotinib as above at a predetermined dose.
  patients requiring surgery were treated 7 days prior to tumor removal; PK analysis and effects of erlotinib on epidermal growth factor receptor (EGFR)
  erlotinib hydrochloride given orally
  Other: pharmacological study, laboratory biomarker analysis.
Arm/Group | Phase 1 Dose Escalation | Phase 2 Recurrent Malignant Gliomas and Nonprogressive Gbm
Serious Adverse Events (participants affected / at risk) | 0/32 | 2/99
Other Adverse Events (participants affected / at risk) | 27/32 | 11/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation (N=32) | Phase 2 Recurrent Malignant Gliomas and Nonprogressive Gbm (N=99)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation (N=32) | Phase 2 Recurrent Malignant Gliomas and Nonprogressive Gbm (N=99)
rash (Skin and subcutaneous tissue disorders) | 19 (19) | 11 (11)
granulocytopenia (Investigations) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 9 (9) | 2 (2)
fatigue (General disorders) | 5 (5) | 3 (3)
nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less